CLINICAL TRIAL: NCT00287391
Title: The Impact of Gastroesophageal Reflux Disease in Sleep Disorders: A Pilot Investigation of Rabeprazole, 20 mg Twice Daily for the Relief of GERD-Related Insomnia.
Brief Title: Sleep Disorders and Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLEEP
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Insomnia; GERD
Keywords: Insomnia; Gastroesophageal Reflux Disease (GERD); Sleep Disturbance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Gastroesophageal Reflux; Parasomnias | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rabeprazole

SUMMARY:
This study will investigate Gastroesophageal Reflux Disease (GERD)as a cause of sleep disturbance. Patients with GERD may experience all or some of the following symptoms: stomach acid or partially digested food re-entering the esophagus (which is sometimes referred to as heartburn or regurgitation) and belching. Even very small, unnoticeable amounts of rising stomach acid may cause patients to wake up during the night.

This study will also investigate the effect of Rabeprazole, (brand name Aciphex) on patients with known insomnia. Rabeprazole is an FDA approved medication already marketed for the treatment of GERD.

DETAILED DESCRIPTION:
Participants with known insomnia will undergo an overnight pH and sleep study. Those found to be eligible after the first sleep study (those with significantly poor sleep quality and no significant sleep apnea) will be started on 2 weeks 20 mgs, twice-a-day, rabeprazole. Upon completion of the 2 week course of rabeprazole, subjects will repeat the overnight pH and sleep studies. Upon completion of these studies, participation is complete.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking male or female subjects, 18-75 years of age. (Women must be two (2) years post-menopausal or surgically sterile. Women of childbearing potential or <1 year post-menopausal must be practicing an approved method of contraception and have a negative urine pregnancy test at screening.),
2. a six-month duration of insomnia,
3. sleep difficulty at least 3 nights per week, and a sleep study demonstrating > 10 arousals/hour for those aged < 45, and >15 for those who are 45 or older.

Exclusion Criteria:

1. BMI > 30 or history of snoring (in order to decrease the prevalence of sleep apnea in the sample),
2. use of any proton pump inhibitor or H2 receptor antagonist within one week of undergoing initial sleep study,
3. previous acid-suppressing medication for sleep disturbances,
4. previous surgical antireflux procedure,
5. current medical therapy that includes digoxin or ketoconazole,
6. previous aerodigestive malignancy,
7. a previously diagnosed psychological or medical cause of insomnia (other than suspected GERD), and
8. inability or unwillingness to provide consent for the procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The percentage of: subjects with non-OSA sleep disturbances who demonstrate esophageal reflux, night-time arousals which are accompanied by a reflux event.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, MPH, Principal Investigator — UNC Gastroenterology
Locations (1):
- UNC Gastroenterology and UNC Sleep Disorders Center, Chapel Hill, North Carolina, United States